CLINICAL TRIAL: NCT05967104
Title: The Effect of Sexual Education in Women With Gynecological Cancer Based On The Plissit Model On Awareness And Attitude in Midwifery Students: A Randomised Controlled Study
Brief Title: Sexual Education in Women Based On The Plissit Model On Awareness And Attitude in Midwifery Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Principal Investigator, yasemin hamlacı başkaya, Head of Midwifery Depatment, Sakarya University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 03072023
Record Dates: First submitted 2023-07-13; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Cancer; Educational Problems; Sex Behavior
Keywords: PLISSIT; sexual education; gynecological cancer; sexual attitudes and beliefs
MeSH Terms: conditions — Neoplasms; Sexual Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Training to the intervention group was carried out in 3 sessions of 45 minutes each week, organized by the first author (AD). In each session, training was organized based on the PLISSIT framework.
  Questionnaires (Introductory individual form, Gynecological cancer awareness scale and Sexual Attitudes and Beliefs Scale) were completed by students included in the intervention and control groups at the beginning and one month after the completion of the 3 training sessions.
  Interventions: Other: Education based on the PLISSIT model
- Control group (No Intervention): The students in the control group were not given any training within the scope of the study, and they only had knowledge about gynecological cancers and sexuality, which are included in the course content of gynecological diseases. However, in order to comply with ethical principles, training information was provided online to the control group after the study data collection process was completed.

INTERVENTIONS:
Other: Education based on the PLISSIT model — Training to the intervention group was carried out in 3 sessions of 45 minutes each week, organized by the first author (AD). In each session, training was organized based on the PLISSIT framework.
  Arms: Experimental group

SUMMARY:
In this study, it was aimed to determine the awareness levels and attitudes of the students with the sexual counseling training conducted in line with the PLISSIT model. This experimental (randomized-controlled) study was conducted with midwifery students who agreed to participate in the study and met the inclusion criteria at a state university in western Turkey. As a result of the randomization, there were 38 students in the intervention group and 36 students in the control group. While training based on the PLISSIT framework was given to the intervention group, no training was given to the control group. Data were collected through the Introductory Information Form, the Gynecological Cancer Awareness Scale (GCPS), and the Sexual Attitudes and Beliefs Scale (CTİÖ) before the training and after the completion of the 3 trainings.

DETAILED DESCRIPTION:
Intervention In order to improve the educational content, researchers conducted a literature review on gynecological cancers, sexual problems in gynecological cancer, sexual counseling. The training content was created after the literature review.

Gynecological cancers are malignant diseases of the ovaries, cervix, endometrium, vulva, vagina and fallopian tubes that make up the female reproductive system. GLOBACAN (Global Cancer Observatory) 2020 data show that gynecological cancers rank fourth among the most common types of cancer among women in the world. Gynecological cancers are responsible for more than 100,000 incidences and 32,000 deaths per year. Significant changes are taking place, especially in the area of sexuality. It is known that sexually active gynecological cancer cases often complain of dyspareunia, vaginal dryness, postcoital bleeding, deterioration in sexual arousal, lack of sexual desire, genitopelvic pain. In addition, changes in the female genital organs, such as vaginal stenosis, vaginal dryness, scar formation in the vagina and vaginal atrophy, can lead to sexual dysfunction. Sexual dysfunction is one of the most common and troubling qualities of life issues faced by women with gynecological cancer, but it is rarely discussed among cancer patients, survivors, and health professionals. Therefore, a comprehensive assessment of sexual health from the first visit of patients should be carried out as a routine part of each examination. In this regard, health professionals need to apply resources that will encourage effective, sensitive, communication with patients about sexual health problems. One of the most widely used interventions in the field of assessing and managing sexual problems is the PLISSIT model. The PLISSIT model provides a safe, tolerant and therapeutic environment for the discussion of sexual concerns, encouraging referral to an appropriate specialist as needed. The model consists of four steps to address sexual concerns: Consent, Limited Information, Specific Recommendations, and Intensive Therapy. The first stage of this model is to allow patients to share their thoughts and concerns about their sex life. In the second stage, individuals are informed about their thoughts and concerns about their sex life. In the third stage, patients are given "special recommendations". Specific recommendations should be appropriate to each person's individual needs. At this point, health professionals need to know more about sexuality in order to give patient-specific information. The fourth stage involves the referral of the patient to the relevant specialist. This model enables healthcare professionals to develop effective strategies for addressing sexual concerns. In order for the model to be applied effectively, it is essential that the relevant health professionals are informed about the subject. In this context, it is very important to show health professionals and students studying in the field of health that sexuality is very important in women with gynecological cancer, to raise their awareness in the field and to ensure that their positive attitudes towards sexuality are formed. For this reason, in this study, 3rd-year students of the midwifery department were trained on "sexuality education for women with gynecological cancer" prepared based on the PLISSIT model, and it was examined how the gynecological cancer awareness and sexual attitudes and beliefs of the students were affected.

In this study, it is aimed to determine the effect of sexuality education in line with the PLISSIT model on the gynecological cancer awareness levels of the students and their sexual attitudes and beliefs.

ELIGIBILITY:
Inclusion Criteria:

* Being a midwifery 3rd year student,
* Agree to participate in the study.

Exclusion Criteria:

-Having failed or not taken the "Gynecology" course even though it is a third year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-07-20 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Gynecological cancer awareness scale change | pre-intervention, 1 month after intervention
  Scale; It consists of four sub-dimensions: routine control and awareness of serious disease perception in gynecological cancers, awareness of gynecological cancer risks, awareness of prevention from gynecological cancers and early diagnosis and information awareness in gynecological cancers.
Sexual Attitudes and Beliefs Scale Change | pre-intervention, 1 month after intervention
  high scores from scale items and grand total; It shows that negative beliefs and attitudes towards evaluating the patient's sexuality/providing sexual counseling increase and there are more obstacles in evaluating sexual problems and providing counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Ahsen DEMİRHAN KAYACIK, Study Chair — Sakarya University
Locations (1):
- Sakarya University, Sakarya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Demirhan Kayacik A, Hamlaci Baskaya Y, Ilcioglu K. Effect of Sexual Counseling Training in Gynecological Cancers According to the PLISSIT Model on Midwifery Students' Awareness and Attitude: A Randomized Clinical Trial. Int J Community Based Nurs Midwifery. 2024 Jul 1;12(3):140-149. doi: 10.30476/IJCBNM.2024.100377.2355. eCollection 2024 Jul. PMID 39161865